CLINICAL TRIAL: NCT05181826
Title: Collection of Blood From Healthy Patients, Patients With Benign Disease and Patients With Cancer
Acronym: ELITE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Helio Genomics (Industry)
Responsible Party: Sponsor
Other Study IDs: 001-2018
Record Dates: First submitted 2021-12-17; First posted 2022-01-06 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2023-07

CONDITIONS: Cancer; Liver Cirrhosis; Chronic Hepatitis; Hepatitis B; Hepatitis C; Diabetes; COPD
MeSH Terms: conditions — Neoplasms; Liver Cirrhosis; Hepatitis, Chronic; Hepatitis B; Hepatitis C; Diabetes Mellitus; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

INTERVENTIONS:
Diagnostic Test: Multi-analyte Blood Test — Intend for the qualitative detection of DNA methylation markers for the detection of various types of cancer

SUMMARY:
To acquire blood samples from subjects for various purposes, including: i) determining the sensitivity and specificity of select DNA methylation markers for the detection of various types of cancer, ii) identifying benign conditions that may induce false positive or false negative results, and iii) defining the effects of potential interfering substances, such as chemotherapy drugs.

DETAILED DESCRIPTION:
Whole blood, plasma, and/or serum specimens will be collected from patients with active cancer, patients in cancer remission, patients diagnosed with benign disease, and healthy volunteers. These blood samples will be used to perform various studies to determine the utility of select DNA methylation markers for cancer diagnostic or prognostic indications.

ELIGIBILITY:
Inclusion Criteria:

2.1.1 Age 18 years or older.

2.1.2 A diagnosis of cancer, cancer remission, benign disease (benign tumor, diabetes, liver cirrhosis, chronic hepatitis B or hepatitis C virus infection, Chronic obstructive pulmonary disease, etc.) or apparently healthy volunteers. .

Exclusion Criteria:

2.2.1 Patients that are unwilling or unable to sign the Informed Consent Form will be excluded.

2.2.2 Approximately 50 mL of blood will be drawn from participants within an 8-week period under this protocol. Patients that have already given 50 mL of blood within this time frame will be excluded.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Healthy subjects, subjects diagnosed with active cancer, subjects in cancer remission, and subjects diagnosed with a benign disease will eligible to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2019-05-21 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Independent performance measure of sensitivity and specificity of a multi-analyte blood test | 1 month
  The primary objective is to measure the performance (sensitivity and specificity) the multi-analyte blood Test for the detection of liver cancers in healthy subjects, subjects diagnosed with active cancer, subjects in cancer remission, and subjects diagnosed with a benign disease.

SECONDARY OUTCOMES:
To investigate potential endogenous and exogenous interfering substances of a multi-analyte blood test | 1 Month
  To investigate potential endogenous and exogenous interfering substances of a multi-analyte blood test for the detection of liver cancers within healthy subjects, subjects diagnosed with active cancer, subjects in cancer remission, and subjects diagnosed with a benign disease.
Ascertain Reference Range(s) | 1 Month
  Ascertain reference range determination(s) for select CpG methylation sites
Ascertain Sample Stability | 1 Month
  Sample stability under various shipping conditions

CONTACTS AND LOCATIONS:
Overall Officials: Taggert, Study Director — Helio Health
Locations (7):
- United States (7):
  - Torrance Memorial Physician Network - Cancer Care, Redondo Beach, California
  - Allina Health, Virginia Piper Cancer Institute, Coon Rapids, Minnesota
  - Virginia Piper Cancer Institute Mercy Hospital-Unity Campus, Fridley, Minnesota
  - VPCI Oncology Research, Minneapolis, Minnesota
  - Methodist LeBonheur Healthcare, Memphis, Tennessee
  - Liver Center of Texas, Dallas, Texas
  - Methodist Hospital, Richardson, Texas